CLINICAL TRIAL: NCT02443584
Title: Pharmacogenetic Testing in an Outpatient Population of Patients With Major Depressive Disorder or Depressive Disorder Not Otherwise Specified With Avera Medical Group Clinics
Brief Title: Pharmacogenetic Testing on an Outpatient Population With a Depression Diagnosis
Acronym: PGX-AMG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AIHG-1430-PGxAMG
Record Dates: First submitted 2015-02-06; First posted 2015-05-14 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Major Depressive Disorder
Keywords: depression; pharmacogenetics; pharmacogenomics; major depressive disorder; genetics; anti-depressants
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 4-Week Group (Other): Pharmacogenetic testing released to physician at 4 weeks following enrollment into study
  Interventions: Other: pharmacogenetic testing
- 12-Week Group (Other): Pharmacogenetic testing released to physician at 12 weeks following enrollment into study
  Interventions: Other: pharmacogenetic testing

INTERVENTIONS:
Other: pharmacogenetic testing — pharmacogenetic testing for anti-depressant/anti-psychotic medications

SUMMARY:
This is a randomized, control group design of pharmacogenetic implementation in a mental health population of subjects taking anti-depressants and/or anti-psychotics with a new or current primary or secondary diagnosis of Major Depressive Disorder (MDD) or Depressive Disorder Not Otherwise Specified (DDNOS).

DETAILED DESCRIPTION:
Mental illness affects one in four adults in the United States; approximately 61.5 million Americans experience mental illness in a given year. According to the National Alliance for the Mentally Ill, the impact of serious mental illness costs Americans $193.2 billion in lost earnings per year. In addition, mental illness patients have an increased risk of having chronic medical conditions, leading to increased costs and emergency service utilization for those conditions. In addition to substantial costs, patients with psychiatric illness are difficult to treat. More than two-thirds of patients with depression do not respond to first line therapy. Treatment often involves numerous trials of individual agents and combinations of medications in order to achieve optimal response. Pharmacogenetic testing is being used in more settings to guide treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* Current primary or secondary diagnosis of Major Depressive Disorder or Depressive Disorder Not Otherwise Specified
* Have moderate to severe depression as identified by PHQ-9 scoring of 10 or greater
* Taking or be newly prescribed an anti-depressant or anti-psychotic medication
* Able to provide informed consent

Exclusion Criteria:

* Pregnant or breastfeeding
* Active and/or unstable diagnosis of substance abuse, excluding nicotine
* Primary diagnosis of dementia, bipolar disorder (any type), schizophrenia, schioaffective disorder, or personality disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Clinical outcomes (response to medication following medication recommendation guided by pharmacogenetic testing) | 24 weeks
  response to medication following medication recommendation guided by pharmacogenetic testing

SECONDARY OUTCOMES:
Clinical utility (Utilization by physicians in following medication recommendations guided by pharmacogenetic testing) | 24 weeks
  Utilization by physicians in following medication recommendations guided by pharmacogenetic testing

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Stanley, MD, Principal Investigator — Avera McKennan Hospital & University Health Center
Locations (1):
- Avera McKennan Hospital & University Health Center, Sioux Falls, South Dakota, United States